CLINICAL TRIAL: NCT07269327
Title: A Phase 1, Open Label, Single Dose, Parallel-group Study to Investigate the Pharmacokinetics of the Fixed Combination of 900 IU r-hFSH and 450 IU r-hLH Given as Pergoveris®, Administered Subcutaneously in Pituitary-suppressed Healthy Premenopausal Female Participants of Japanese or Caucasian Origin
Brief Title: An Ethno-bridging Study of Pergoveris in Healthy Premenopausal Participants of Japanese or Caucasian Origin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS132705_0006; 1012476 (Registry Identifier: IRAS)
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Fertility
Keywords: Clinical pharmacology; gonadotropins; infertility; prefilled pen; ethnicity
MeSH Terms: conditions — Infertility | interventions — Desogestrel; Ethinyl Estradiol; pergoveris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Japanese Female Participants (Experimental)
  Interventions: Drug: Desogestrel and ethinylestradiol fixed dose combination; Combination Product: Follitropin alfa/lutropin alfa
- Group 2: Caucasian Female Participants (Experimental)
  Interventions: Drug: Desogestrel and ethinylestradiol fixed dose combination; Combination Product: Follitropin alfa/lutropin alfa

INTERVENTIONS:
Drug: Desogestrel and ethinylestradiol fixed dose combination — Participants will self-administer one tablet of desogestrel and ethinylestradiol fixed dose combination once daily to ensure downregulation.
  Other Names: Marvelon
Combination Product: Follitropin alfa/lutropin alfa — Participants will receive a combination product of follitropin alfa and lutropin alfa subcutaneously (SC) on Day 1 after confirmation of down regulation.
  Other Names: Pergoveris

SUMMARY:
The purpose of this study is to assess the Pharmacokinetic (PK) of Recombinant human follicle-stimulating hormone (follitropin alfa) (r-hFSH) and Recombinant human luteinizing hormone (lutropin alfa) (r-hLH) following a single subcutaneous injection of Pergoveris in pituitary-suppressed healthy female participants of Japanese or Caucasian origin. Study details include:

Study Duration: Approximately 9 weeks Treatment Duration: Approximately 4 weeks downregulation with Marvelon® and a single dose of Pergoveris.

Visit Frequency: Once in the Screening period, twice in the Downregulation period, and 8 continuous days in the study site during the Confinement period.

ELIGIBILITY:
Inclusion Criteria:

* Participant who are overtly healthy, as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participant who have a negative urine pregnancy test before starting Marvelon and on the day before the Pergoveris dose (Day -1)
* Participant who have a normal baseline FSH (< 12 IU/L) and E2 levels less than or equal (<=) 100 picogram per mililiter (pg/mL) and follicles <= 11 millimeter (mm) in diameter at Screening
* Participant who have a normal ThinPrep® cytologic test (TCT) during Screening
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Participant with any condition that, in the Investigator's opinion, constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Participants with any clinically significant abnormalities of the genital organs as determined by gynecological examination and transvaginal ultrasound scan (TVUS) and based on the Investigator's judgment (e.g. ovarian tumors, nonfunctional ovarian cysts, and endometrial hyperplasia)
* Participant with imminent planned major surgery
* Participant with a History of tumors of the pituitary gland or hypothalamus
* Other protocol defined exclusion criteria may apply

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Baseline-Adjusted Area Under the Serum Concentration- Time Curve from Time Zero to Last Quantifiable Sampling Time After Administration (AUC0-tlast,adj) for both r-hFSH and r-hLH | Predose (baseline), 2 hour(hr), 4, 6, 7, 8, 9, 10, 12,15 and 18hr post-dose on Day 1; 24hr, 36hr post-dose on Day 2; 48hr post-dose on Day 3; 72 hr post dose on Day 4; 96hr post-dose on Day 5; 120hr post-dose on Day 6 and 168hr post-dose on Day 8
Baseline- Adjusted Maximum Observed Serum Concentration (Cmax,adj), for both r-hFSH and r-hLH | Predose (baseline), 2 hour(hr), 4, 6, 7, 8, 9, 10, 12,15 and 18hr post-dose on Day 1; 24hr, 36hr post-dose on Day 2; 48hr post-dose on Day 3; 72 hr post dose on Day 4; 96hr post-dose on Day 5; 120hr post-dose on Day 6 and 168hr post-dose on Day 8

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs | From Screening to End of Study (approximately 9 weeks)
Number of Participants with Clinically Significant Change From Baseline in Laboratory Parameters | Baseline (Day -1) upto end of study (approximately 9 weeks)
  The laboratory assessment includes biochemistry, coagulation, hematology, hormonal, urinalysis parameters.
Number of Participants With Abnormal Vital Signs | Up to end of study (Approximately 9 Weeks)
  Vital signs included body temperature, systolic and diastolic blood pressure, respiratory rate and pulse rate and electrocardiogram (ECG) measurements.
Participants Serum Estradiol (E2) levels | Screening (Day -53 to Day -24) and Day-1
Number of Participants With Abnormal Follicle Size and Number measured by Transvaginal Ultrasound (TVUS) | Day-2 to Day-1 (Downregulation), and Day 6 to Day 8
Number of Participants Experiencing Local Reactions | Baseline up to end of study (approximately 9 weeks)
  Pain, redness, swelling, bruising, and itching around the injection site will be assessed.
Serum Concentration of Baseline- Adjusted r-hFSH and r-hLH | Predose (baseline), 2 hour(hr), 4, 6, 7, 8, 9, 10, 12,15 and 18hr post-dose on Day 1; 24hr, 36hr post-dose on Day 2; 48hr post-dose on Day 3; 72 hr post dose on Day 4; 96hr post-dose on Day 5; 120hr post-dose on Day 6 and 168hr post-dose on Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Fortrea Clinical Research Unit Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html